CLINICAL TRIAL: NCT04909983
Title: A Single Center Explorative Study of the Treamtent ofDiabetes Patients With Contact Dermatitits Caused byInsulin Infusion Pump or Glucose Monitor
Brief Title: An Explorative Study of Treatment of Contact Dermatitis Due to DiabetesDevices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped after 17/20 participants due to lack of time after a prolonged recrutiment period.
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Anna Korsgaard Berg, Principal Investigator MD, Copenhagen University Hospital at Herlev
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPLX-PT01
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Contact Dermatitis Irritant; Type 1 Diabetes
MeSH Terms: conditions — Dermatitis, Irritant; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Medical Device, an occlusive patch for 3 days.
  Interventions: Device: DPLX-PT1
- Control (Active Comparator): Standard of Care
  Interventions: Other: Control arm

INTERVENTIONS:
Device: DPLX-PT1 — A polymer skin patch for occlusional therapy
  Arms: Intervention
Other: Control arm — Standard of care
  Arms: Control

SUMMARY:
A feasibility study of treatment with a occlusive medical device or patch in pediatric patients with type 1 diabetes suffering from irritative contact dermatitis due to diabetes devices.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, and for patients under the legal age consent by a legal guardian
* Clinically confirmed, active and evaluable irritant contact dermatitis (ICD)
* Age 6-20 at the time of signing the informed consent form (ICF)
* Ability to answer study questionnaires

Exclusion Criteria:

* Any type of skin irritation other than ICD
* Use of occlusive therapy for the treatment of their ICD, or unwilling to refrain from this treatment for duration of study
* For any other reason considered unsuitable by the investigator
* Pregnant or of child-bearing potential unwilling to use acceptable effective contraception

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Response rate of active treatment versus standard of care | 8 days after active treatment compared to 8 days after standard of care

SECONDARY OUTCOMES:
Time to resolution of Irritative contact dermatitis | After 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Anna Korsgaard Berg, MD, Principal Investigator — Pediatric Department, Herlev Hospital
Locations (1):
- Pediatric Department, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No